CLINICAL TRIAL: NCT06250907
Title: Evaluation of Accuracy of Implant Placement for Patients With Mandibular Reconstruction Using Dynamic Navigation Compared to Static Guides: a Parallel, Randomized Controlled Clinical Trial
Brief Title: Accuracy of Implant Placement for Patients With Mandibular Reconstruction Using Dynamic Navigation and Static Guides
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDC-24-2
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-11

CONDITIONS: Mandibular Deficiency
MeSH Terms: conditions — Micrognathism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic navigation (Experimental)
  Interventions: Procedure: The guidance of dynamic navigation
- Static template (Active Comparator)
  Interventions: Procedure: The guidance of static template

INTERVENTIONS:
Procedure: The guidance of dynamic navigation — Osteotomy and implant placement with the guidance of dynamic navigation
  Arms: Dynamic navigation
Procedure: The guidance of static template — Osteotomy and implant placement with the guidance of static template
  Arms: Static template

SUMMARY:
To evaluate and compare the accuracy of implant placement using dynamic navigation technique versus static template technique in patients with bone tissue flap reconstruction of mandibular defects, thus further guiding the clinical application of dynamic navigation systems to assist in conventional implant placement in patients with mandibular defects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 18 and 70 (inclusive)
* Mandibular defects (including Class I defects, limited to the body of the mandible; Class II defects, muscular-mandibular region defects and Class III defects, chin protrusion-muscular-mandibular region defects), which have been reconstructed by mandibular vascularization of free iliac bone, and fibular composite muscular flap grafts for greater than 3 months
* Normal mouth opening (≥ 40 mm)
* Trialists voluntarily signed an informed consent form before performing any research-related experimental steps.

Exclusion Criteria:

* Presence of localized inflammation in adjacent teeth, including uncontrolled periodontitis (periodontal probing to a depth of >4 mm)
* Presence of untreated acute and chronic apical periodontitis in adjacent teeth
* Oral mucosal lesions (e.g., lichen planus)
* Adjacent teeth with space-occupying lesions (including cysts, tumors, etc.)
* Systemic diseases affecting bone healing, wound healing and dental implant treatment (e.g., uncontrolled diabetes mellitus, fasting blood glucose ≥ 8.8 mmol/L despite medication)
* Uncontrolled and unstabilized severe hypertension
* Contraindications to routine implant surgery and oral surgery
* Heart disease (Class II or above)
* Patients with liver or kidney insufficiency or abnormality
* Obese patients with body mass index (BMI) > 28 kg/m2
* Patients with a history of full-dose radiotherapy, localized radiotherapy to the head or neck
* Patients requiring long-term high-dose steroid therapy
* Patients who are receiving or have received in the last 3 months medications (e.g., bisphosphonates) that may affect or promote bone metabolism
* Consecutive antibiotic therapy or chronic anti-inflammatory therapy (≥3 times per week) within the first 4 weeks of starting the procedure
* Alcohol or chronic substance abuse
* Immunocompromised patients
* Smoking/tobacco equivalents/chewing tobacco >10 cigarettes per day
* Physical or mental impairment that interferes with the performance of oral hygiene care
* Female patients who are pregnant or breastfeeding
* Patients who, in the opinion of the investigator, have poor compliance and cannot participate in the trial
* Patients who have participated in a clinical trial of another drug or device within 30 days prior to the start of the procedure (Study Day 0)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-29 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Three-dimensional implant placement accuracy of apical point | Postoperative day 2±1
  The postoperative cone beam computed tomography (CBCT) was aligned to the preoperative plan in specific software, and the three-dimensional coordinates of the preoperatively planned and actual postoperative implant placement positions were measured separately, from which the three-dimensional distance (in mm) between the apical point of the actual implant and the apical point of the virtual implant was calculated.

SECONDARY OUTCOMES:
Three-dimensional implant placement accuracy of coronal point | Postoperative day 2±1
  The postoperative CBCT was aligned to the preoperative plan in specific software, and the three-dimensional coordinates of the preoperatively planned and actual postoperative implant placement positions were measured separately, from which the three-dimensional distance (in mm) between the coronal point of the actual implant and the coronal point of the virtual implant was calculated.
Three-dimensional implant placement angular accuracy | Postoperative day 2±1
  The postoperative CBCT was aligned to the preoperative implant placement plan in specific software to measure the three-dimensional coordinates of the preoperative plan and the actual postoperative implant placement position, respectively, and to calculate the angle (°) between the actual implant and the mid-axis of the virtual implant accordingly.
Operation time | Intraoperative
  From the beginning of anesthesia to the complete removal of the static template or navigation reference frame.
Patient subjective satisfaction | Postoperative day 14±1
  Evaluating patient satisfaction with the visual analogue scale
Failure rate during implant healing period | Postoperative day 90±7
  1. According to the definition of Albrektsson and Zarb in 1986, the healing period is considered successful if the following conditions are met: no loosening of the implant after removal of the upper restoration; no peri-implant radiolucency; no peri-implant bone instability; and no pain. Implant retention was evaluated according to three levels: good osseointegration, poor osseointegration, and implant failure. 2. Implant survival rate = (N total - N failure)/(N total) × 100%.